CLINICAL TRIAL: NCT07110415
Title: A Randomized Controlled Trial of the Efficacy and Safety of Yangxinshi Tablets in the Treatment of Patients With Coronary Heart Disease Complicated by Cardiac Dysfunction
Brief Title: Efficacy and Safety Trials of Yangxinshi Tablets in the Treatment of Patients With Coronary Heart Disease Complicated by Cardiac Dysfunction
Acronym: HEARTPOWER
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: SPH Qingdao Growful Pharmacetical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Growful2401YXS
Record Dates: First submitted 2025-07-22; First posted 2025-08-07 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Coronary Heart Disease; Cardiac Dysfunction
Keywords: Yangxinshi; Coronary heart disease; Cardiac dysfunction
MeSH Terms: conditions — Coronary Disease | interventions — Yangxinshi

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial group (Experimental): Basic treatment and Trial drug
  Interventions: Drug: Yangxinshi tablet
- Control group (Sham Comparator): Basic treatment
  Interventions: Drug: Blank control

INTERVENTIONS:
Drug: Yangxinshi tablet — Basic treatment: All patients received a conventional treatment regimen, including outcome-improving drugs (aspirin, P2Y12 receptor inhibitor、β-blockers, statins, ARNI /ACEI/ARB, SGLT2i, and MRA) and symptom-relieving drugs (nitrates, calcium antagonists, and loop diuretic).
  Trial drug: Yangxinshi tablets, 3 tablets/3 times a day, taken orally
  Other Names: Yangxinshi
  Arms: Trial group
Drug: Blank control — Basic treatment: All patients received a conventional treatment regimen, including outcome-improving drugs (aspirin, P2Y12 receptor inhibitor、β-blockers, statins, ARNI /ACEI/ARB, SGLT2i, and MRA) and symptom-relieving drugs (nitrates, calcium antagonists, and loop diuretic).
  Trial drug: Blank control
  Arms: Control group

SUMMARY:
A randomized controlled trial was conducted to evaluate the efficacy and safety of Yangxinshi tablets in improving the condition of patients with coronary heart disease complicated by cardiac dysfunction.

DETAILED DESCRIPTION:
The purpose of this study was to investigate whether the addition of Yangxinshi tablets to conventional treatment can reduce the composite endpoint time, increase exercise tolerance, and improve quality of life and mental health in patients with coronary heart disease complicated by cardiac dysfunction. A total of 2708 eligible patients were randomly divided into two groups. In addition to conventional treatment, the trial group was given Yangxinshi tablets (3 tablets/time, 3 times/day), while the control group was a blank control. The treatment cycle continued until the expected number of endpoint events was reached or the study ended, whichever occurred first. The primary endpoint was the composite endpoint of ischemic events or heart failure-related clinical events (including all-cause death, ischemia-driven revascularization, stroke, myocardial infarction (MI), and readmission due to aggravated ACS or heart failure) during the study period.

ELIGIBILITY:
Inclusion Criteria:

1. For inpatients diagnosed with coronary heart disease (including acute coronary syndrome and chronic coronary syndrome), it is up to the doctor to decide whether to undergo revascularization and what kind of revascularization to use.
2. Patients aged between 40 and 80 years (inclusive), regardless of sex;
3. Patients with NYHA cardiac function classes II-IV;
4. Patients with NT-proBNP > 125 pg/mL (or BNP>35 pg/mL);
5. The syndrome differentiation in traditional Chinese medicine conforms to chest obstruction (qi deficiency and blood stasis syndrome)
6. Patients who voluntarily participated and signed an informed consent form.

Exclusion Criteria:

1. Patients with STEMI within 3 days;
2. Patients at extremely high risk of NSTEMI (hemodynamic instability, cardiogenic shock, new-onset heart failure or aggravated heart failure, severe ventricular arrhythmia)
3. Patients with acute myocardial infarction complicated with cardiogenic shock, mechanical complications, respiratory failure and other multiple organ failure;
4. Patients with severe liver dysfunction (transaminase levels more than three times the upper limit of normal), renal insufficiency (eGFR < 30mL/min/1.73m2), acute infectious diseases, and mental disorders;以上翻译结果来自有道神经网络翻译（YNMT）· 通用场景
5. Patients with drug-resistant hypertension (systolic blood pressure ≥180 mmHg and/or diastolic blood pressure ≥110 mmHg);
6. Pregnant or lactating women, or those planning pregnancy during the study period;
7. Patients who cannot tolerate 3 months of dual antiplatelet therapy;
8. Patients with allergic reactions or abnormal drug reactions to the study drug or any of its excipients;
9. Patients who have regularly taken Yangxinshi tablets and similar traditional Chinese medicine, Chinese patent medicine or traditional Chinese medicine decoction with the same curative effectin the past month;
10. Patients who have participated in other clinical drug trials within the last three months;
11. Patients with malignant tumors and other pathological conditions with an expected survival of less than 3 years;
12. Patients whom the investigator deems unsuitable for participating in the clinical trial.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2708 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2030-08-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
The composite endpoint was ischemic events or heart failure-related clinical events | Through study completion, an average of 3 years
  All-cause death, ischemia-driven revascularization, stroke, MI, and readmission due to aggravated ACS or heart failure

SECONDARY OUTCOMES:
Ischemic composite endpoint events | Through study completion, an average of 3 years
  Cardiovascular and cerebrovascular death, MI, ischemia-driven revascularization, stroke, and readmission due to ACS
Heart failure-related clinical events | Through study completion, an average of 3 years
  Readmission due to aggravated heart failure or all-cause death
Cardiovascular and cerebrovascular deaths | Through study completion, an average of 3 years
  Occurrence of cardiovascular and cerebrovascular deaths
All-cause death | Through study completion, an average of 3 years
  Occurrence of all-cause death
Readmission due to ACS | Through study completion, an average of 3 years
  Readmission due to ACS
Readmission due to aggravated heart failure | Through study completion, an average of 3 years
  Readmission due to aggravated heart failure
The cumulative incidence of readmission due to aggravated ACS or heart failure | Through study completion, an average of 3 years
  The joint gamma frailty model was adopted for analysis
Win ratio | Through study completion, an average of 3 years
  The main efficacy indicators were analyzed by using the win ratio method
6MWD | From baseline at 48 weeks
  Change in 6-minute walking distance
NT-proBNP or BNP | From baseline at 48 weeks
  Measurement of NT-proBNP or BNP, calculation of the proportion of patients achieving NT-proBNP <125 pg/mL (or BNP <35 pg/mL), and the degree of reduction
Patient Health Questionnaire - 9(PHQ-9) depression scale | After 24 and 48 weeks of treatment
  The Patient Health Questionnaire - 9(PHQ-9)depression scale comprises nine questions. In each assessment area, scores range from 0 to 3 based on the increasing frequency of difficult: 0 indicates "not at all," 1 indicates "sometimes," 2 indicates "more than half the time," and 3 indicates "almost every day." The total score ranges from 0 to 27,higher scores mean a worse outcome.
Generalized Anxiety Disorder 7 - item Scale(GAD-7) anxiety scale | After 24 and 48 weeks of treatment
  The Generalized Anxiety Disorder 7 - item Scale(GAD-7) anxiety scale comprises seven questions. In each assessment area, scores range from 0 to 3 based on the increasing frequency of difficult: 0 indicates "not at all," 1 indicates "sometimes," 2 indicates "more than half the time," and 3 indicates "almost every day." The total score ranges from 0 to 21,higher scores mean a worse outcome.
NYHA | After 24 and 48 weeks of treatment
  Changes in New York Heart Association (NYHA) functional classification
SAQ | After 24 and 48 weeks of treatment
  Changes in Seattle Angina Questionnaire (SAQ) scores.The SAQ scale is divided into 5 dimensions, with a total of 19 items, and each item is scored out of 100 points. The higher the score, the better the therapeutic effect
KCCQ-OS | After 24 and 48 weeks of treatment
  Changes in Kansas City Cardiomyopathy Questionnaire overall score (KCCQ-OS) compared to baseline.The total score ranges from 0 to 100,higher scores mean a better outcome.
Echocardiography | After 48 weeks of treatment
  Changes from baseline examined via echocardiography, including left ventricular systolic function (left ventricular end-diastolic diameter (LVDd), left ventricular end-systolic diameter (LVSd), left ventricular ejection fraction (LVEF), left ventricular fractional shortening (FS) and left ventricular diastolic function (E/A and E/e) . When possible, the left ventricular global longitudinal strain rate (LVGLS) was also measured
Metabolic equivalents(METs) | After 48 weeks of treatment
  Changes in metabolic equivalents(METs) determined by cardiopulmonary exercise testing in some patients.
Anaerobic thresholds (ATs) | After 48 weeks of treatment
  Changes in anaerobic thresholds (ATs) determined by cardiopulmonary exercise testing in some patients.
Maximal oxygen consumption (VO2max) | After 48 weeks of treatment
  Changes in maximal oxygen consumption (VO2max) determined by cardiopulmonary exercise testing in some patients.
VO2/heart rate(HR) | After 48 weeks of treatment
  Changes in VO2/HR determined by cardiopulmonary exercise testing in some patients.
The ratio of the change in VO2 to the change in the work rate (△VO2/△WR) | After 48 weeks of treatment
  Changes in △VO2/△WR determined by cardiopulmonary exercise testing in some patients.

OTHER OUTCOMES:
Heart rate | After 24 and 48 weeks of treatment
  Unit: beats /minute
Blood pressure | After 24 and 48 weeks of treatment
  Systolic and diastolic,unit: mmHg
12-lead Electrocardiogram (ECG) | After 24 and 48 weeks of treatment
  12-lead ECG consists of Ⅰ、Ⅱ、Ⅲ、aVR、aVL、aVF、V1、V2、V3、V4、V5、V6.ECG consists of P wave, PR interval, QRS complex, ST segment, and T wave.
White blood cell (WBC) count | After 24 and 48 weeks of treatment
  Normal value: 4-10, unit: 109/L.Check at 24 and 48 weeks to see if it is within the normal range.
Red blood cell (RBC) count | After 24 and 48 weeks of treatment
  Normal value: 3.5-5, unit: 1012/L.Check at 24 and 48 weeks to see if it is within the normal range.
Hemoglobin (Hb) level | After 24 and 48 weeks of treatment
  Normal value: 110-150, unit: g/L.Check at 24 and 48 weeks to see if it is within the normal range.
Platelet (PLT) count | After 24 and 48 weeks of treatment
  Normal value: 100-300,unit: 109/L.Check at 24 and 48 weeks to see if it is within the normal range.
Liver function test | After 24 and 48 weeks of treatment
  Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)
Serum creatinine concentration | After 24 and 48 weeks of treatment
  Unit: μmol /L
Estimated glomerular filtration rate (eGFR) | After 24 and 48 weeks of treatment
  Unit: ml/minute.Calculated using the Modification of Diet in Renal Disease (MDRD) equation
Adverse events | Through study completion, an average of 3 years
  Adverse events/serious adverse events

CONTACTS AND LOCATIONS:
Locations (96):
- China (96):
  - The People's Hospital of Bozhou, Haozhou, Anhui
  - Beijing Hospital of Traditional Chinese Medicine, Beijing, Beijing Municipality
  - Dongfang Hospital,Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - Guang'anmen Hospital,China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Army Specialty Medical Center, Chongqing, Chongqing Municipality
  - Chongqing Emergency Medical Center, Chongqing, Chongqing Municipality
  - Chongqing General Hospital, Chongqing, Chongqing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - The Southwest Hospital of Amu, Chongqing, Chongqing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - The affiliated traditional Chinese medicine hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The first affiliated hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - The Fifth Affiliated Hospital,Sun Yat-sen University, Zhuhai, Guangdong
  - The First Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The First Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The First Affiliated Hospital of Zunyi Medical University", Zunyi, Guizhou
  - Baoding No.1 Central Hospital, Baoding, Hebei
  - Jingjiang People's Hospital, Cangzhou, Hebei
  - Handan Central Hospital, Handan, Hebei
  - Hebei General Hospital, Shijiazhuang, Hebei
  - Xingtai People's Hospital, Xingtai, Hebei
  - The First Affiliated Hospital of Hebei North University, Zhangjiakou, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - The First Affiliated Hospital of Harbin Medical University, Haerbin, Heilongjiang
  - The Second Affiliated Hospital of Harbin Medical University, Haerbin, Heilongjiang
  - HeGang People's Hospital, Hegang, Heilongjiang
  - Mudanjiang Cardiovascular Disease Hospital, Mudanjiang, Heilongjiang
  - The 7th People's Hospital of Zhengzhou, Zhengzhou, Henan
  - The Third People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Hunan Provincial TCM Hospital, Changsha, Hunan
  - Yiyang Central Hospital, Yiyang, Hunan
  - Xuyi People's Hospital, Huai'an, Jiangsu
  - Nanjing Lishui People's Hospital, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Jiangsu Provincial People's Hospital Suqian Branch, Suqian, Jiangsu
  - Taizhou Fourth People's Hospital, Taizhou, Jiangsu
  - Xuzhou No.1 People's Hospital, Xuzhou, Jiangsu
  - Affiliated Hospital of Changchun University of Traditional Chinese Medicine, Changchun, Jilin
  - Jilin Provincial People's Hospital, Changchun, Jilin
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - The Second Norman Bethune Hospital of Jilin University, Changchun, Jilin
  - Jilin People's Hospital, Jilin, Jilin
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Dandong Central Hospital, Dandong, Liaoning
  - Fushun Central Hospital, Fushun, Liaoning
  - Fuxin Central Hospital, Fuxin, Liaoning
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The Fourth Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Chifeng Municipal Hospital, Chifeng, Neimenggu
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong University of Traditional Chinese Medicine Affiliated Hospital, Jinan, Shandong
  - The 960th Hospital of the PLA Joint Logistics Support Force, Jinan, Shandong
  - The Fourth People's Hospital of Jinan, Jinan, Shandong
  - The Second People's Hospital of Liaocheng, Liaocheng, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Tengzhou Central People's Hospital, Tengzhou, Shandong
  - Affiliated Hospital of Shandong Second Medical University, Weifang, Shandong
  - PLA Joint Logistics Support Force No.970 Hospital, Yantai, Shandong
  - Yantai Affiliated Hospital of Binzhou Medical University, Yantai, Shandong
  - Fudan University Minhang Hospital, Shanghai, Shanghai Municipality
  - Ruijin Hospital Luban Branch, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Songjiang Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Xi'an Gaoling District Hospital, Xi’an, Shanxi
  - The Eighth Affiliated Hospital,Sun Yat-sen University, Shenzhen, Shenzhen
  - Chengdu Wenjiang District People's Hospital, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Guang'an People's Hospital, Guang’an, Sichuan
  - The People's Hospital of Jianyang City, Jiancheng, Sichuan
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - Tianjin Fifth Center Hospital, Tianjin, Tianjin Municipality
  - Tianjin Hospital of Integrated Traditional Chinese and Western Medicine, Tianjin, Tianjin Municipality
  - Yunnan Provincial Hospital of Traditional Chinese Medicine, Kunming, Yunnan
  - Affiliated Hangzhou First People's Hospital,School of Medicine,Westlake University, Hangzhou, Zhejiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - The First Hospital of Jiaxing, Jiaxing, Zhejiang
  - The Second Hospital of Jiaxing, Jiaxing, Zhejiang
  - Beilun Branch of the First Affiliated Hospital of Zhejiang University School of Medicine, Ningbo, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang
  - The Affiliated People'sHospital of Ningbo University, Ningbo, Zhejiang
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Shaoxing, Zhejiang
  - Taizhou Central Hospital, Taizhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - Yantai Yuhuangding Hospital, Yantai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vrints C, Andreotti F, Koskinas KC, Rossello X, Adamo M, Ainslie J, Banning AP, Budaj A, Buechel RR, Chiariello GA, Chieffo A, Christodorescu RM, Deaton C, Doenst T, Jones HW, Kunadian V, Mehilli J, Milojevic M, Piek JJ, Pugliese F, Rubboli A, Semb AG, Senior R, Ten Berg JM, Van Belle E, Van Craenenbroeck EM, Vidal-Perez R, Winther S; ESC Scientific Document Group. 2024 ESC Guidelines for the management of chronic coronary syndromes. Eur Heart J. 2024 Sep 29;45(36):3415-3537. doi: 10.1093/eurheartj/ehae177. No abstract available. PMID 39210710
- [Result] Li Y, Li Y, Zhang Z, Zhang J, Chen H, Yu H, Meng X, Yuan H, Shao L, Lu Y, Liu B, Xu J, Zhang Y, Li J, Han Y; HEARTRIP investigators. Efficacy and safety of yangxinshi versus trimetazidine on exercise tolerance in patients with coronary heart disease after percutaneous coronary intervention: Multicenter, double-blind clinical trial. Phytomedicine. 2024 Dec;135:156198. doi: 10.1016/j.phymed.2024.156198. Epub 2024 Nov 7. PMID 39566404
- [Result] Zhang S, Shen Y, Liu P, Meng X, Hu D. Yangxinshi Tablet Improves Exercise Capacity for Patients with Coronary Heart Disease: Results from a Randomized, Double-Blind, Placebo-Controlled, and Multicenter Trial. Rev Cardiovasc Med. 2022 Jul 21;23(8):266. doi: 10.31083/j.rcm2308266. eCollection 2022 Aug. PMID 39076617
- [Result] Rao SV, O'Donoghue ML, Ruel M, Rab T, Tamis-Holland JE, Alexander JH, Baber U, Baker H, Cohen MG, Cruz-Ruiz M, Davis LL, de Lemos JA, DeWald TA, Elgendy IY, Feldman DN, Goyal A, Isiadinso I, Menon V, Morrow DA, Mukherjee D, Platz E, Promes SB, Sandner S, Sandoval Y, Schunder R, Shah B, Stopyra JP, Talbot AW, Taub PR, Williams MS; Peer Review Committee Members. 2025 ACC/AHA/ACEP/NAEMSP/SCAI Guideline for the Management of Patients With Acute Coronary Syndromes: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. J Am Coll Cardiol. 2025 Jun 10;85(22):2135-2237. doi: 10.1016/j.jacc.2024.11.009. Epub 2025 Feb 27. PMID 40013746